CLINICAL TRIAL: NCT05407233
Title: Interdisciplinary Care for the Patient With Type 2 Diabetes: Promoting Improvement in the Quality of Care at an Outpatient Level and Seeking Answers to Clinical Practice Questions - Reuse of Inputs and Placebo Intervention Effects
Brief Title: Reusing Needles for Subcutaneous Insulin Injection in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-0574
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Reuse needle; Insulin administration
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be carried out to compare the reuse or not of needles in diabetes patients who use insulin. The groups will be divided in two: a group that will not reuse the needles and a group that will reuse the needles five times. Primary outcomes as skin complications, local pain, glycemic control will be evaluated at baseline and after 4, 8 and 12 weeks and secondary outcomes will also be evaluated as quality of life, insulin application technique, frequency of capillary blood glucose tests, adherence to treatment, quality of needles, microbiological contamination and cost-utility analysis of after needle reuse
Who Masked: Outcomes Assessor
Masking Description: The study was blinded to the professionals involved in the analyses of skin complications and the needle characterization test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Doesn´t reuse the syringe for insulin application
  Interventions: Device: Does not reuse the syringe for insulin application
- Group 2 (Experimental): Uses the syringe five times to insulin application
  Interventions: Device: Uses the syringe for insulin delivery five times

INTERVENTIONS:
Device: Does not reuse the syringe for insulin application — Does not reuse needles for insulin application Patients will be given quantity of needles for use during the study period according to the allocated group and a collector for sharps descarpack to collect the used syringes and needles. Initially, all patients will be instructed on the indication and importance of insulin use, aspects of conservation, preparation and administration, reviewing the dose aspirated in the syringe. They will also be instructed in relation to the use of the collector for sharps. Patients will also receive the booklet specially designed for this registry where they must indicate the number of hematomas, bruises, lipodystrophies, or inflammation that they identify whenever they occur. This booklet will be given to the team of researchers at each visit (monthly), who will review the records with the patient and guide them for subsequent completion.
  Arms: Group 1
Device: Uses the syringe for insulin delivery five times — Uses the needles for insulin application five times. Patients will be given quantity of needles for use during the study period according to the allocated group and a collector for sharps descarpack to collect the used syringes and needles. Initially, all patients will be instructed on the indication and importance of insulin use, aspects of conservation, preparation and administration, reviewing the dose aspirated in the syringe. They will also be instructed in relation to the use of the collector for sharps. Patients will also receive the booklet specially designed for this registry where they must indicate the number of hematomas, lipodystrophies, or inflammation that they identify whenever they occur. This booklet will be given to the team of researchers at each visit (monthly), and they will review the records with the patient and guide them for subsequent completion.
  Arms: Group 2

SUMMARY:
A randomized clinical trial (RCT) will be carried out to compare the reuse or not of needles in patients with type 2 diabetes (T2DM) that use insulin. Two groups will be studied: a group that will not reuse the needles and a group that will reuse the needles five times. The aim of this study is to evaluate related outcomes such as bruises, infection, lipodystrophy, pain and glycemic control, whether or not to reuse insulin delivery needles in patients with T2DM who use insulin.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a highly prevalent chronic disease with increasing incidence worldwide. It is well demonstrated in the literature that adequate glycemic control can reduce the incidence of chronic complications. The Brazilian Ministry of Health must provide patients with diabetes with the necessary resources for optimal glycemic control. However, this supply is often not enough and the population ends up reusing needles and lancets. According to the Brazilian National Health Surveillance Agency (ANVISA) and the manufacturers, it is recommended to use the needle for insulin application only once, but a report from the Brazilian Society of Diabetes shows that half of the patients disregard this rule - some reuse each needle up to five times. Studies show that patients do not like carrying extra needles when they are away from home, are reluctant to carry containers to dispose used needles, and decide that it is not worthwhile worth buying a new needle for each injection. Others describe that injections from reused needles are not noticeably more painful as long as they do not reuse them excessively. Finally, some patients believe that disposing of a needle after use is ecologically wasteful because metal and plastic must be incinerated. A randomized clinical trial will be carried out to compare the reuse or not of needles in patients with diabetes who use insulin. Primary outcomes as skin complications, local pain, glycemic control will be evaluated at baseline and after 4, 8 and 12 weeks and secondary outcomes will also be evaluated as quality of life, insulin application technique, frequency of capillary blood glucose tests, adherence to treatment, quality of needles, microbiological contamination and cost-utility analysis of after needle reuse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM
* Over 18 years of age
* Reuses each syringe at least three times for insulin application.

Exclusion Criteria:

* Use of insulin pens
* Pregnant women
* Patients undergoing chemotherapy
* Use of anticoagulants
* Clotting disorders, lesions or skin changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Change in glycemic control | Baseline and Month 3
  For assessment of glycemic control, HbA1c will be requested if the patient has not performed the test in the last month at the initial meeting and at the end of the study, after 12 weeks, for all patients.
Change in Skin complications | Baseline, Month1, Month 2 and Month 3
  Dermatological conditions will be evaluated for the formation of hematomas, ecchymoses, appearance of lipodystrophy (lipohypertrophy and lipoatrophy), signs of inflammation and pain in the applications. In the follow-up meetings, the skin complications presented by the patient at the insulin injection sites will be recorded through photography by the professional. To aid in the evaluation of skin complications, a partnership will be established carried out with the TeleHealth Program, where distance and standard pixel size will be used for photos of patients' skin complications through a professional digital camera.
Change in Pain assessment | Baseline, Month1, Month 2 and Month 3
  The evaluation of pain in the application of insulin will be evaluated through a one-dimensional numerical scale of pain intensity, according to the clinical record in the follow-up meetings which consists of numbers from 0 to 10 (0 = " no pain" to 10= "worst pain imaginable").

SECONDARY OUTCOMES:
Evaluate the quality of needles after reuse of the insulin administration needle compared to non-reuse. | Month 2
  Needle quality evaluation will be performed through the penetration test and drag through using the Mecmesin digital dynamometer (Advanced Force Gauge).
Evaluate the microbiological contamination after reuse of the insulin administration needle compared to non-reuse. | Month 2
  To evaluate the microbiological contamination of the needles, the semi-quantitative culture method of the external surface of the needle will be carried out (Maki's method).
Insulin Injection technique | Baseline and Month 3
  The iInsulin Injection technique will be evaluated through the Insulin Injection Technique Questionnaire (ITQ) which consists of an initial session with the patient, followed by observation of the injection technique and examination of the injection sites by the researcher.
Adherence to diabetes treatment | Baseline, Month1, Month 2 and Month 3
  Adherence to treatment will be verified using the SCI-R questionnaire (Self Care Inventory- Revised Version), validated for Portuguese. Is a 15-item questionnaire, on a 5-point Likert scale that reflects how well the subjects followed recommendations for self-care during the past month (1 = "never" to 5 = "always").
Quality of life assessment | Baseline, Month1, Month 2 and Month 3
  The quality of life with a focus on insulin application will be evaluated through the DQOL-Brazil questionnaire (Diabetes Quality Of Life Measure). DQOL consists of 4 domains (satisfaction, impact, social/vocational worries, and diabetes-related worries) whose answers are scored from 1 to 5. Lower scores indicate higher quality of life. The "social/vocational worries" domain was excluded because most of our participants were retired or inactive.
Frequency of capillary blood glucose tests | Baseline
  Information related to capillary blood glucose monitoring of included patients and other information such as ways of acquiring supplies.
Frequency of reuse of lancets of included patients | Baseline
  Information related to capillary blood glucose monitoring of included patients and other information such reuse of lancets will be evaluated by completing a form at the initial meeting.
Analyze cost-utility | Baseline, Month1, Month 2 and Month 3
  Costs will be estimated from several standard cost lists. The survey of costs will be based on the values of sale sold in the Brazilian market and in accordance with the table of procedures of the Unified Health System (SUS). Outcomes will be evaluated using a health outcome unit that combines gain (or loss) in survival with quality of life, the unit is the quality-adjusted life year (quality adjusted life year, QALY).

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Agord Schaan, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Gabriela Berlanda, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No